CLINICAL TRIAL: NCT06349538
Title: Identifying Markers of Disease Subtypes and Disease Progression in the Syndrome of Essential Tremor - a Prospective Cohort Study
Brief Title: Identifying Markers of Disease Subtypes and Disease Progression in the Syndrome of Essential Tremor
Status: Enrolling by invitation | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: 35-435 ex 22/23
Record Dates: First submitted 2024-03-28; First posted 2024-04-05 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Essential Tremor
Keywords: essential tremor; subtypes; neurodegeneration; biomarkers; MRI; imaging; sGFAP; sNfL; tremor analysis
MeSH Terms: conditions — Essential Tremor; Nerve Degeneration | interventions — Physical Examination; Blood Specimen Collection; Ultrasonography; Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Essential tremor patients: Essential tremor patients will undergo a detailed clinical examination incl. motor/non motor scoring systems and questionnaires, blood draw, sonography, tremor analysis and cerebral MRI. Additionally, essential tremor patients will undergo optic coherence tomography and olfcatory mucosa swab for alpha-synuclein.
  All tests are conducted at baseline as well as at a follow-up examination 5 years later.
  No drugs or other interventions are to be administered
  Interventions: Diagnostic Test: Clinical examination, blood draw, cerebral MRI, sonography, tremor analysis, OCT, olfactory mucosa swab.

INTERVENTIONS:
Diagnostic Test: Clinical examination, blood draw, cerebral MRI, sonography, tremor analysis, OCT, olfactory mucosa swab. — see previous descriptions

SUMMARY:
The goal of this observational study is to learn about epidemiology, biologic markers, disease subtypes and possible prognostic factors in essential tremor (ET) patients. The main question[s] it aims to answer are:

* The prevalence of ET-plus compared to ET in a prospectively collected ET population.
* To assess in detail the heterogenous group of ET patients using comprehensive clinical (motor and non-motor scales, questionnaires), imaging [magnetic resonance imaging (MRI), sonography of substantia nigra and cerebral vessels], neurophysiological (tremor analysis, digital spiral drawing) and laboratory markers (sGFAP, sNfL, routine laboratory parameters).
* To assess possible non-invasive markers of neurodegeneration in ET patients (optic coherence tomography, alpha-synuclein in olfactory mucosa)

Participants will be asked to undergo the above mention evaluation at baseline and at follow-up approx. 5 years later.

Researchers will compare the findings within the ET group to independently existing cohorts of healthy controls and/or patients with other movement disorders like Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Presence of an essential tremor syndrome according to MDS consensus criteria or suspected incipient essential tremor (differential diagnosis vs. enhanced physiological tremor)
* Patient is able and willing to give informed consent.
* age above 18 years.

Exclusion Criteria:

* Patient is not able or not willing to give informed consent.
* Existence of a legal representative.
* age below 18 years

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: ET-patients will be recruited from all patients visiting a tertiary neurological hospital and its various institutions (emergency department, outpatient clinic, specialised outpatient clinic for movement disorders, ward patients) for any neurologic complaint.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2034-04-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of ET-plus | approx. 2 years
  Determine the prevalence of ET-plus within a prospectively collected ET population

SECONDARY OUTCOMES:
Age of ET patients | 1 minute; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  age at disease onset and age at baseline
Sex of ET patients | 1 minute; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  male, female, other
Family history | 1 minute; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  positive or negative for essential tremor or Parkinson's disease
Symptom leading to ET-plus classification | 1 minute; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  e.g. rest tremor, impaired tandem gait, mild parkinsonian signs, questionable dystonia, mild cognitive impairment
current and former medication for essential tremor | 2 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  e.g. propranolol yes vs no, topiramate yes vs no, primidone yes vs no
subjective disease course of ET | 1 minute; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  no progression, slowly and continuously, relapsing, plateau-like after initial progression, rapidly progressive
responsivity to alcohol | 1 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  amelioration of tremor severity after consumption of alcohol (yes vs. no vs. unknown)
presence of cardiovascular risk factors | 2 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  arterial hypertension yes vs. no, hyperlipidemia yes vs. no, smoking yes vs. no vs. former, diabetes mellitus yes vs. no, coronary artery disease yes vs. no
MDS-UPDRS (Movement Disorder Society Unified Parkinson's Disease Rating Scale) parts I-IV | 20-30 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  rates clinical severity of parkinsonian symptoms, range 0-260 points with higher points meaning more severe symptoms
modified Essential Tremor Rating Assessment Scale (mTETRAS) | 10 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  rates clinical severity of ET symptoms, ranging from 0-80 (the "modified" means the inclusion of 2 additional items rating rest tremor) with higher points meaning more severe motor symptoms; also includes a subscale rating activities of daily living ranging from 0-48 points with more points meaning more severe disability due to ET
Scale for the assessment and rating of ataxia (SARA) | 5-10 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  assesses symptoms of ataxia, ranging from 0 (no ataxia) to 40 (most severe ataxia)
Verbal fluency animals (part of the CERAD-plus test battery) | 1 minute; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  patients needs to say as many animals as possible within 1 minute, the more, the better
Boston Naming Test (part of the CERAD-plus test battery) | 2 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  the patient needs to name 15 items (shown as pictures) correctly, the more, the better
Mini Mental State Examination Test (MMSE; part of the CERAD-plus test battery) | 3-5 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  a cognitive screening test with a minimum of 0 and a maximum of 30 points
word list learning (part of the CERAD-plus test battery) | 10 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  the patient is shown 10 words which he needs to remember and repeat immediately after reading them (within 90 seconds); there a three tries; the more he remembers, the better
constructive praxis (part of the CERAD-plus test battery) | 20-30 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  the patient needs to draw 4 figures from a model which are then rated according to prespecified criteria (maximum of 11 points, the more the better)
word list recall (part of the CERAD-plus test battery) | 90 seconds; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  the patient needs to remember as many of the 10 words learned in "word list learning"; time limit 90 seconds
word list recognition (part of the CERAD-plus test battery) | 2 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  the patient needs decide whether a word shown to him was part of the 10 words learned before; there a 20 words in total, and 10 each were part of the learned words while 10 where not; the more he/she remembers correctly, the better (1 point for each correctly identified word)
constructive praxis recall (part of the CERAD-plus test battery) | 3-4 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  the patients needs to draw the 4 figures from "constructive praxis" from memory; they are then rated according to the same criteria with a maximum of 11 points
Trail Making Test A (part of the CERAD-plus test battery) | 2 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  the patient needs to connect numbers in ascending order from 1 to 25, time is measured in seconds (the faster, the better)
Trail Making Test B (part of the CERAD-plus test battery) | 2 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  the patient needs to connect numbers and letters in ascending and alternating order from 1 to 13 and A to L, respectively, time is measured in seconds (the faster, the better)
s-words (part of the CERAD-plus test battery) | 1 minute; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  the patient needs to list as many words starting with the letter "s" within 60 seconds as possible; the more the better
Frontal Assessment Battery (FAB) | 5 - 10 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  a neuropsychological test focusing on executive function, ranging from 0 (most impaired) to 18 (normal)
Geriatric Depression Scale (GDS) | 3-5 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  a short questionnaire rating depressive symptoms, ranging from 0 (no depressive symptoms) to 15 (most severe depressive symptoms)
Hospital Anxiety and Depression Scale (HADS) | 5 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  a questionnaire rating anxiety and depressive symptoms, ranging from 0 (no depressive/anxious symptoms) to 42 (most severe symptoms)
Non-Motor Symptoms Scale for Parkinson's Disease (NMSS) | 5 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  a questionnaire rating non motor symptoms, ranging from 0 (no symptoms) to 128 (most severe non motor symptoms)
RBD Screening Questionnaire | 2 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  rates probability for the presence of RBD (REM sleep behavior disorder) using 13 questions; points are given from 0 to 13 with higher points indicating a higher probability for RBD
Global Physical Activity Questionnaire (GPAQ) | 5-7 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  the GPAQ is a questionnaire provided by the WHO and rates the extent of physical (-in-) activity; rating is done according to the WHO manual available from the WHO website
Quality of Life in Essential Tremor Questionnaire (QUEST) | 5 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  a questionnaire rating quality of life specifically in ET patients; ranging from 0 (best quality of life) to 120 points (worst quality of life)
University of Pennsylvania Smell Identification Test (UPSIT) | 10-15 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  a smell test ranging from 0 (worst olfactory function) to 40 points (best olfactory function)
Montreal Cognitive Assessment (MOCA) | 5-10 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  a screening cognitive test rating cognitive dysfunction from 0 (worst) to 30 (best)
Auditory verbal learning test | 5 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  assesses how well patients can remember 15 words after hearing them; the more they can remember, the better
Symbol Digit Modalities Test (SDMT) | 90 seconds; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  patients need to translate specific symbols into numbers (1-9) using a key; they more the can translate in 90 seconds, the better
Brief Visuospatial Memory Test | 2-3 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  patients can look at 6 figures for 10 seconds each, then they have to reproduce them; 3 trials; the more they remember, the better
Comprehensive trail making test 4 | 1-2 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  patients have to connect numbers (1 to 21) in ascending order with lines; time is measured in seconds; the faster, the better
Comprehensive trail making test 5 | 1-2 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  patients have to connect numbers (1 to 13) and letters (A to L) in ascending order and alternatingly with lines; time is measured in seconds; the faster, the better
Regensburg word fluency test | 2 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  patients have to list words starting with "g" or "r" alternatingly or things within the categories of "clothes" or "flowers" alternatingly; they have 1 minute for each of the two tasks, the more they can list, the better
EQ-5D | 1-2 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  a quick questionnaire (5 questions) rating quality of life, ranging from 0 (very bad) to 1 (best)
resilience scale (RS-13) | 1-2 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  a quick questionnaire rating resilience, ranging from 13 (least resilience) to 91 points (highest resilience)
Pittsburgh Sleep Quality Index (PSQI) | 3-4 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  a quick questionnaire rating sleep quality, ranging from 0 (best sleep) to 21 points (worst sleep quality)
Digital Spiral Drawing | 2-3 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  patients are asked to draw Archimedes spirals (a total of 4, 2 with each hand) on a standard tablet PC using a touchpen; the process is done using a free available website-based application (http://www.trsper.com/); the main outcome is visual rating of the spirals ranging from 0 (perfectly normal) to 9 (worst spiral)
Schellong Test | 3.5 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  blood pressure test for orthostatic hypotension; blood pressure is measured non-invasively using a automatic device at the left arm in seating position and after 1 and 3 minutes of standing; orthostatic hypotension is defined as a drop in systolic blood pressure of 20mmHg or more and/or of diastolic blood pressure of 10mmHg or more
serum glial fibrillary acidic protein (sGFAP) | 5 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  sGFAP-level is measured from serum using SIMOA-technology
serum neurofilament light (sNfL) | 5 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  sNfL-level is measured from serum using SIMOA-technology
Transcranial sonography | 10 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  the presence of hyperechogenicity (yes/no and area in cm2) of the substantia nigra is measured using transcranial sonography
tremor analysis | 20 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  tremor frequency and total tremor power are measured
cerebral MRI | 45 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  white matter hyperintensities (volume in mm3)
cerebral MRI | 45 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  presence of lacunes (number of)
cerebral MRI | 45 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  cerebral microbleeds (number of)
cerebral MRI | 45 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  volumetry of total brain and regions (in mm3)
cerebral MRI | 45 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  Diffusion tensor imaging parameters (fractional anisotropy, mean diffusivity, radial diffusivity)
cerebral MRI | 45 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  nigrosome-1-imaging (presence of swallow tail sign yes vs. no)
optic coherence tomography (OCT) | 5-10 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  thickness of retinal nerve fiber layer in both eyes and each quadrant and in vicinity of the macula and papilla
optic coherence tomography (OCT) | 5-10 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  thickness of ganglion cell layer in both eyes and each quadrant and in vicinity of the macula and papilla
optic coherence tomography (OCT) | 5-10 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  thickness of inner plexiform layer in both eyes and each quadrant and in vicinity of the macula and papilla
optic coherence tomography (OCT) | 5-10 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  thickness of choroidea in both eyes and each quadrant and in vicinity of the macula and papilla
Olfactory mucosa swab | 5-10 minutes; Baseline (recruiting time approx. 2 years) and follow-up (5 years after individual baseline)
  swab of the olfactory mucosa testing for alpha-synuclein using a seeding assay (outcome: presence of misfolded alpha-synuclein yes vs. no)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Austria, Austria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bhatia KP, Bain P, Bajaj N, Elble RJ, Hallett M, Louis ED, Raethjen J, Stamelou M, Testa CM, Deuschl G; Tremor Task Force of the International Parkinson and Movement Disorder Society. Consensus Statement on the classification of tremors. from the task force on tremor of the International Parkinson and Movement Disorder Society. Mov Disord. 2018 Jan;33(1):75-87. doi: 10.1002/mds.27121. Epub 2017 Nov 30. PMID 29193359
- [Background] Doustar J, Torbati T, Black KL, Koronyo Y, Koronyo-Hamaoui M. Optical Coherence Tomography in Alzheimer's Disease and Other Neurodegenerative Diseases. Front Neurol. 2017 Dec 19;8:701. doi: 10.3389/fneur.2017.00701. eCollection 2017. PMID 29312125
- [Background] Stefani A, Iranzo A, Holzknecht E, Perra D, Bongianni M, Gaig C, Heim B, Serradell M, Sacchetto L, Garrido A, Capaldi S, Sanchez-Gomez A, Cecchini MP, Mariotto S, Ferrari S, Fiorini M, Schmutzhard J, Cocchiara P, Vilaseca I, Brozzetti L, Monaco S, Jose Marti M, Seppi K, Tolosa E, Santamaria J, Hogl B, Poewe W, Zanusso G; SINBAR (Sleep Innsbruck Barcelona) group. Alpha-synuclein seeds in olfactory mucosa of patients with isolated REM sleep behaviour disorder. Brain. 2021 May 7;144(4):1118-1126. doi: 10.1093/brain/awab005. PMID 33855335